CLINICAL TRIAL: NCT03261258
Title: ICU and Contact Person: Comparison of Criteria for Designation in Patients and Close Friends and Relatives
Brief Title: Comparison of Criteria for the Designation of a Contact Person in ICU Patients and Close Friends and Relatives
Acronym: REPERE II/III
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: QUENOT 2016
Record Dates: First submitted 2017-08-23; First posted 2017-08-24 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Patients Hospitalised in a Medical ICU
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Patients hospitalised in the ICU of Dijon CHU Burgundy
  Interventions: Other: Questionnaire
- Proches: Relatives/close friends of patients hospitalised in the ICU of Dijon CHU Burgundy
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire

SUMMARY:
In the vast majority of cases, the person of trust (or contact person) is not designated by the patient (emergency, severe disease situations, coma, sedation, etc.). The healthcare team thus identifies a person who 1) may not be the person the patient would have designated and 2) may not be the most suitable to take on this responsibility. Though the first point is not easy, the main difficulty for the clinician is to know if he is dealing with the "right person for the job", meaning a person who is able to take on the responsibility of the contact person. This is a heavy responsibility in terms of the information given, of passing on this information to relatives and friends, of consulting the doctors, of help or support in medical decisions, etc. This responsibility may also be difficult for one person alone to take on and it may be helpful to share it between several friends or relatives. In a princeps study (QUENOT, 2015), it was shown that the process used by the healthcare team to designate a contact person was based on criteria such as knowledge of the wishes and values of the patient, the strength of the relationship with the patient, and the person of trust designated before admission to the ICU. However, we do not know what criteria are used by the patients themselves or those used by their close friends and relatives. This study will make it possible to determine and to measure the possible differences between the criteria used by the ICU healthcare team (REPERE I), those used by patients (REPERE III) and finally, those used by close friends and relatives (REPERE II).

In order to do this, 300 persons (150 patients and 150 relatives/friends) will complete questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Patients and their friends/relatives who have been given information on the study
* Patients admitted to the ICU according to the criteria defined by decree n° 2002-465 of the law of 5 April 2002 relative to the rights of patients and the quality of the healthcare system;
* Patients unable to designate a person of trust on admission;
* Patients able to designate a person of trust on discharge from the ICU.

Exclusion Criteria:

* Refusal to participate;
* Age < 18 years;
* Patient/relative under ward of court;
* Patient/relative presenting a major cognitive disorder ruling out a reliable interview;
* Patient and/or relative who cannot be interviewed or who cannot provide information ;
* Absence of family and/or close friends.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the medical ICU of Dijon CHU Burgundy and their relatives/friends.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Difference between scores measured (relatives/patients) on the scales for the principal criteria for the designation of a contact person | at baseline

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France

REFERENCES:
- [Result] Rigaud JP, Hardy JB, Meunier-Beillard N, Devilliers H, Ecarnot F, Quesnel C, Gelinotte S, Declercq PL, Eraldi JP, Bougerol F, Quenot JP. The concept of a surrogate is ill adapted to intensive care: Criteria for recognizing a reference person. J Crit Care. 2016 Apr;32:89-92. doi: 10.1016/j.jcrc.2015.12.011. Epub 2015 Dec 21. PMID 26787167